CLINICAL TRIAL: NCT02387203
Title: Clinical Trial to Define the Effect of Perioperative H. Pylori Eradication With Antibiotic Treatment on Long Term Outcomes of Patients With Pseudomyxoma Peritonei of Appendiceal Origin Undergoing Cytoreductive Surgery/Hyperthermic Intraperitoneal Chemotherapy
Brief Title: Antibiotic Treatment and Long-term Outcomes of Patients With Pseudomyxoma Peritonei of Appendiceal Origin
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Mercy Medical Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MMC-2014-53
Record Dates: First submitted 2015-01-19; First posted 2015-03-12 (Estimated); Last update posted 2024-11-19 (Actual); Status verified 2024-11

CONDITIONS: Pseudomyxoma Peritonei; Appendiceal Neoplasms
Keywords: Pseudomyxoma Peritonei; Appendiceal cancer; CRS/HIPEC; PMP
MeSH Terms: conditions — Pseudomyxoma Peritonei; Appendiceal Neoplasms | interventions — Lansoprazole; Amoxicillin; Clarithromycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PrevPac (Experimental): Study intervention: PrevPac (Prevacid, Amoxicillin, Clarithromycin)twice daily x 14 days for 2 courses (preoperative and post-operative).
  All eligible patients with a PMP diagnosis, undergoing CRS/HIPEC treatment, who consent to study participation will have a urea breath test prior to the first course of PrevPac.
  After surgery, when tolerated, each patient will take a second course of PrevPac. Patients will be seen for follow-up as clinically indicated until year 5.
  Interventions: Drug: PrevPac (Prevacid, Amoxicillin, Clarithromycin)
- PMP Historical Control (No Intervention): The historical control group will consist of all PMP patients who did not receive perioperative antibiotic treatment.

INTERVENTIONS:
Drug: PrevPac (Prevacid, Amoxicillin, Clarithromycin) — 30mg Prevacid, 1g amoxicillin, 500mg clarithromycin administered together for oral use, twice daily for 14 days preoperatively and twice daily for 14 days at least 4 weeks postoperatively
  Other Names: PREVPAC, U.S. Patent No. 5,013,743
  Arms: PrevPac

SUMMARY:
The purpose of this study is to determine the impact of antibiotic therapy on the disease progression and overall survival of patients with Pseudomyxoma Peritonei (PMP).

DETAILED DESCRIPTION:
Single center, open label, historical controlled, phase II study that proposes two courses of standard H. Pylori eradication antibiotic therapy can suppress carcinogenesis and improve the long-term outcomes of patients with PMP. The first course of antibiotics (PrevPac) will be administered before cytoreductive surgery and HIPEC and the second course afterwards. The historical control group will consist of all PMP patients from Mercy Medical Center's Tumor Registry who did not receive perioperative antibiotic treatment. Long-term statistical outcomes will be calculated using the Kaplan-Meier method and Cox proportional hazard ratio to compare pertinent variable. 80 subjects to be enrolled over 2 years, with a 5 year follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have measurable pseudomyxoma peritonei from appendiceal origin, confirmed by histology, cytology, or radiographical evidence -
* Age ≥ 21 years
* Eastern Cooperative Oncology Group (ECOG) performance status score≤2/Karnofsky performance status of (KPS) ≥ 70% (see Appendix B)
* Patients must have normal organ and marrow function as defined below:

Absolute neutrophil count (ANC) ≥1,000/mm3 Platelets ≥100,000/mm3 Hemoglobin ≥ 8.5 g/dL

Renal function:

Creatinine ≤1.5 times the upper limit of normal (ULN) or calculated creatinine clearance ≥60ml/min

Hepatic function:

Bilirubin ≤1.5 times ULN Alanine aminotransferase (ALT) ≤3 times ULN Aspartate aminotransferase (AST) ≤3 times ULN

* Ability of subject or Legally Authorized Representative (LAR) to understand and willingness to sign a written informed consent, approved by Mercy Medical Center Institutional Review Board (IRB)
* A negative pregnancy test for women of childbearing age with all reproductive organs intact

Exclusion Criteria:

* Patients receiving any other investigational agents
* Presence of other invasive malignancies or evidence of another cancer present within the last 3 years, excluding skin cancer
* history of, or known allergic reaction/hypersensitivity to PREVPAC or any component of similar chemical or biologic composition to PREVPAC
* Patients < 21 of age
* Pregnancy or lactation at the time of proposed assignment. Pregnant women are excluded from this study because PREVPAC is based on the pregnancy category for clarithromycin which is Category C agent with the potential for teratogenic or abortifacient effects. These potential risks may also apply to CRS/HIPEC.
* Assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol (e.g., unable to swallow pills)
* Psychiatric or addictive disorders or other conditions that, in the opinion of the investigator, would preclude the patient from meeting the study requirements or giving informed consent
* Known active acute hepatitis and confirmed diagnosis of Human Immunodeficiency Virus (HIV) infection. HIV-positive patients on combination antiretroviral therapy are ineligible. These patients are at increased risk of lethal infections when treated with marrow-suppressive therapy.
* Active systemic infection that requires use of parenteral antibiotics
* Renal insufficiency with serum creatinine level ≥1.5 times the upper limit of normal or calculated -
* Patients with concurrent severe medical problems unrelated to malignancy that will preclude compliance with the study or places at an unacceptable risk for participation in the study determinate by study investigators
* Patients to be maintained on any medication having severe interactions with PREVPAC

Min Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2015-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5 year
  Kaplan-Meier survival estimates

SECONDARY OUTCOMES:
Progression-free survival measured by no evidence of disease progression, i.e. tumor markers within normal limits, no radiographical evidence of disease | 5 year
  Kaplan-Meier survival estimates

OTHER OUTCOMES:
Tolerance and safety of PrevPac administration | Through 14 day treatment therapy
  Rate of morbidity and mortality
Analyze number of live bacteria in PMP tumor and mucin | through study completion, an average of 5 years
  In situ hybridization [ISH], either bright light or fluorescence in situ hybridization [FISH]

CONTACTS AND LOCATIONS:
Overall Officials: Armando Sardi, M.D., Principal Investigator — Mercy Medical Center; Scott Merrell, PhD, Principal Investigator — Uniformed Sciences University, Health Sciences
Locations (1):
- Mercy Medical Center, Baltimore, Maryland, United States